CLINICAL TRIAL: NCT04852640
Title: Mitigating the Impact of Shoulder Movement Dysfunction; a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PMR-2021-29615
Record Dates: First submitted 2021-04-14; First posted 2021-04-21 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Shoulder Injuries; Shoulder Pain
MeSH Terms: conditions — Shoulder Injuries; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Rehabilitation Program (ARP) (Experimental): Participants will be treated for symptomatic shoulder instability with the evidence-based, targeted treatment intervention. For eight weeks, there will be two treatment sessions per week lasting 30-45 minutes. Exercises in the ARP include: Low-load and high-duration rotator cuff strengthening exercises, progressive scapular muscle endurance training, plyometric strengthening exercises, and surface electromyographic (EMG) biofeedback. Each prescribed exercise in the ARP will be increased to match the participant's function at the discretion of the study clinician. Although the components of the ARP will be pre-determined, the parameters and volumes of the components will be determined and documented over the treatment phase.
  Interventions: Procedure: Active Rehabilitation Program (ARP)
- Nonspecific Passive Intervention (NPI) (Experimental): Participants will be treated for symptomatic shoulder instability with the non-specific, generalized treatment intervention. For eight weeks, there will be two treatment sessions per week lasting 30-45 minutes. The NPI consists of a general approach to treating shoulder pain with passive modalities for pain modulation. These interventions are commonly practiced but have little evidence to support their use in the treatment of symptomatic shoulder instability. Although the components of the NPI will be pre-determined, the parameters and volumes of the components will be determined and documented by a study clinician over the treatment phase.
  Interventions: Procedure: Nonspecific Passive Intervention (NPI)

INTERVENTIONS:
Procedure: Active Rehabilitation Program (ARP) — The ARP intervention consists of therapeutic exercises designed to increase shoulder strength and endurance using a cluster of common exercises used for the treatment of shoulder pain. Specifically, the ARP program will focus on increasing scapular motor-control through a phasic program of common therapeutic exercises. This concept has been shown in the literature as capable of reducing shoulder pain and improving function in a variety of pathological conditions, however, the effect of this approach to reducing pain and increasing function for symptomatic shoulder instability is unknown. The selection of exercises and application for each exercise included in the ARP is based on recommendations from the literature and will incorporate participant feedback to customize dosages.
  Arms: Active Rehabilitation Program (ARP)
Procedure: Nonspecific Passive Intervention (NPI) — The NPI intervention consists of a non-specific treatment approach to shoulder pain that is commonly administered in the clinical setting. Specifically, passive modalities such as ultrasound, massage, and sensory electric stimulation are commonly prescribed in the treatment of shoulder pain to modulate pain. Further, general core strengthening exercises are often implemented. Therefore, the NPI will consist of regularly prescribed passive treatments and general core strengthening exercises, as commonly administered in routine treatment of shoulder pain.
  Arms: Nonspecific Passive Intervention (NPI)

SUMMARY:
The purpose of the proposed work is to screen the effectiveness of an evidence-based, targeted, treatment intervention versus a non-specific, generalized, treatment intervention to treat symptomatic shoulder instability in collegiate swimmers. The results of the study will allow direct observation of treatment effects designed to mitigate the effects of symptomatic shoulder instability. These results will facilitate the optimization of future treatments and interventions.

DETAILED DESCRIPTION:
Currently, there is an unmet need for an effective method to treat shoulder instability. Namely, there is minimal evidence to mitigate the impact of shoulder instability with non-surgical interventions. The presence of shoulder instability can drastically decrease upper extremity function and lead to subsequent shoulder pathology. While there is observational and retrospective evidence to support the use of specific, guided, therapeutic exercise interventions to treat shoulder instability, there are only two randomized controlled trials (RCT) investigating the effects of these types of interventions. While current evidence demonstrates that rehabilitation interventions are capable of decreasing pain and improving self-reported function in individuals with MDI, these investigations include heterogeneous samples and lack thorough investigation of the biomechanical effects of these interventions. The results of this study will allow direct observation of treatment effects designed to mitigate the effects of symptomatic shoulder instability with gold-standard biomechanical techniques. These results will facilitate the optimization of future treatments and interventions. Further, the results will contribute to the current field of musculoskeletal medicine by enhancing biomechanics-based treatment interventions and promote patient-reported outcomes research. The long-term goal of the proposed research is to expand to investigations of treatment effectiveness to more diverse populations and a broader range of movement-related shoulder dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Be an active member of the University of Minnesota Intercollegiate swim team
* Be able to actively raise arm over 150 degrees as measured with a standard goniometer

Exclusion Criteria:

* Are pregnant or are trying to get pregnant
* Are breastfeeding
* Have a previous history of shoulder surgery within the past 12 months
* Have neck pain at the time of enrollment
* Do not speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Change in the magnitude of humeral head translations relative to the scapular glenoid | Within four weeks of treatment initiation and within four weeks of treatment termination
  The magnitude of humeral head translations will be measured as the distance traveled by the humeral head relative to the scapular glenoid. The units of measure for this variable is distance, recorded in millimeters (mm). These measurements will be recorded with biplane radiographic motion analysis.
Change in the magnitude of 3D scapular rotations | Within four weeks of treatment initiation and within four weeks of treatment termination
  The magnitude of 3D scapular rotations will be measured as scapular rotations in each anatomical plane relative to the thorax. The three scapular rotations that will be measured are: scapular upward/downward rotation, scapular internal/external rotation, and scapular anterior/posterior tilting. These rotations are measured in degrees. These measurements will be recorded with biplane radiographic motion analysis.
Changes in average visual analog scale (VAS) | Ten minutes to complete; Weekly for nine months, within 1 week of the intervention initiation, within 1 week of the intervention termination, and eight weeks after intervention
  Pain ratings will be measured with a 10cm VAS. The VAS will not have numbers on the scale, as a numeric pain scale would have. Participants will report their pain rating on the VAS scale weekly by sliding the marker along the line on the electronic survey throughout the duration of the study.
Change in Western Ontario Instability Index (WOSI) | Ten minutes to complete; Weekly for nine months, within 1 week of the intervention initiation, within 1 week of the intervention termination, and eight weeks after intervention
  The WOSI contains 21 items, each rated on a scale of 0 to 100, and four overarching groups: physical symptoms, sports/recreation/work, lifestyle, and emotion. Composite scores range from 0-2100, where greater scores indicate a reduced quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Staker, PhD, PT, Principal Investigator — University of Minnesota Medical School Department of Rehabilitation Medicine
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No